CLINICAL TRIAL: NCT01590537
Title: Prospective Multicentre Non-interventional Comparative Study of Long-term Intrauterine Contraceptives Acceptability and User Satisfaction
Brief Title: Non-interventional Study of Long-term Intrauterine Contraceptives Acceptability and User Satisfaction
Acronym: Mirabel
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15508; MA1010RU (Other: company internal)
Record Dates: First submitted 2012-05-02; First posted 2012-05-03 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Contraception
Keywords: non-interventional; Mirena; Contraception; Russian Federation
MeSH Terms: interventions — Levonorgestrel; Intrauterine Devices, Copper

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Drug: Levonorgestrel (Mirena, BAY86-5028)
- Group 2
  Interventions: Device: Copper IUD

INTERVENTIONS:
Drug: Levonorgestrel (Mirena, BAY86-5028) — intrauterine system containing 52 mg levonorgestrel, with daily release of 20 mcg levonorgestrel
  Groups: Group 1
Device: Copper IUD — Copper device, inserted intrauterine
  Groups: Group 2

SUMMARY:
This is local prospective, non-interventional multi-center comparative study. Primary study objective is evaluation of the user satisfaction with Mirena or Copper IUD up to 1 year after insertion ( patient assessment questionnaire) in daily practice. For each patient, the treating gynecologist documents demographics, medical data, safety parameters and treatment signs and symptoms at an initial visit and one or two follow-up visit(s).

ELIGIBILITY:
Inclusion Criteria:

* Women 20-40 years old
* Parity ≥ 1 child
* Requesting long-term contraception
* Written informed consent.

Exclusion Criteria:

* in accordance with the current leaflet

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females who plan long-term contraception and meet criteria of inclusion and exclusion.
Sampling Method: Non-Probability Sample
Enrollment: 2348 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
User satisfaction of the contraception method with Mirena or Copper IUD | up to 12 months

SECONDARY OUTCOMES:
Safety evaluation of Mirena or Copper IUD in routine practice Safety parameters include number of AEs, severity,relationship to Mirena or Cooper IUD | up to 12 months
Contraceptive reliability of Mirena or Cooper IUD in routine practice ( fixing number of pregnancies) | up to 12 months
Continuation/discontinuation rate ( number of cases with contraceptive method continuation and discontinuations) | up to 12 months
Relationship between different parameters and women preferences in choosing Mirena or Cooper IUD as their contraceptive method ( demographic parameters, age group, residence, reproductive history and plans, etc.) using patients questionnaire | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Russia